CLINICAL TRIAL: NCT02434523
Title: Double-blind Placebo Controlled Trial of the Treatment of Chronic Laryngitis With Amitryptiline
Brief Title: Trial of the Treatment of Chronic Laryngitis With Amitryptiline
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: concern regarding study design
Sponsor: Boston Medical Center (Other)
Collaborators: American Laryngological Association (Other)
Responsible Party: Principal Investigator, J Pieter Noordzij, BMC Attending Physician, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-29925
Record Dates: First submitted 2015-04-22; First posted 2015-05-05 (Estimated); Results first posted 2016-11-30 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-10

CONDITIONS: Laryngeal Diseases; Chronic Laryngeal Neuropathy
Keywords: laryngeal sensory neuropathy
MeSH Terms: conditions — Laryngeal Diseases | interventions — Amitriptyline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- amitriptyline (Experimental): Subjects in this arm will receive pills composed of amitryptline and Avicel (cellulose filler)
  Interventions: Drug: Amitriptyline
- Placebo (Placebo Comparator): Subjects in this arm will receive pills composed only of Avicel (cellulose filler)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Amitriptyline — Subjects in this arm will receive pills composed of amitryptline and Avicel (cellulose filler), starting at 12.5mg nightly, and allowed to increase daily dose by 12.5mg with each subsequent week after enrollment if symptoms not resolved and no adverse effect noted at prior dose, up to maximum dose of 50mg nightly. Treatment duration is 8 weeks
  Other Names: treatment arm
  Arms: amitriptyline
Other: Placebo — Subjects in this arm will receive pills composed of only Avicel (cellulose filler), starting at 12.5mg nightly, and allowed to increase daily dose by 12.5mg with each subsequent week after enrollment if symptoms not resolved and no adverse effect noted at prior dose, up to maximum dose of 50mg nightly. Treatment duration is 8 weeks
  Other Names: placebo arm
  Arms: Placebo

SUMMARY:
The study will compare the effectiveness of amitriptyline versus placebo (inactive medication) in treating chronic laryngitis.

DETAILED DESCRIPTION:
The study will compare the effectiveness of amitriptyline versus placebo (inactive medication) in treating chronic laryngitis. At the baseline visit, subjects will be assigned at random to amitriptyline or placebo which they will take for 8 weeks. Subjects will be seen in the clinic at baseline and at 8 weeks. Improvement will be measured using standardized symptom scales, and a self-reported subjective improvement percentage.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older and able to consent for themselves.
* Structural pathology such as tumor previously ruled out using flexible laryngoscopy.
* Able to speak and read the English language.
* Failed a trial of a proton pump inhibitor for the treatment of gastopharyngeal reflux.
* Women under 55 years of age who may become pregnant must have a negative pregnancy test and agree to barrier or hormonal methods of contraception during the study.

Exclusion Criteria:

* Environmental allergies.
* Smoking within past 5 years.
* Using ginko bilboa (or unwilling to cease using it).
* Current upper respiratory infections.
* Use of narcotics (e.g. oxycodone, methadone).
* Any prior history of amitryptiline use.
* Use of monoamine oxidase inhibitors (MAOIs) within the past 4 weeks (selegiline, phenelzine, tranylcypromine, isocarboxazid, rasagiline, phenelzine sulfate, selegiline hydrochloride, rasagiline mesylate, tranylcypromine sulfate).
* History of urinary retention.
* Any history of major depressive disorder.
* Any prior history of allergy to a tricyclic antidepressant.
* Current diagnosis of gastroesophageal reflux (GERD).
* For women 18-55 years of age without history of menopause: currently nursing or pregnant, plans to become pregnant, or unwillingness to utilize contraception (barrier or hormonal methods).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Pieter Noordzij, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
No plan to share individual data. Data in aggregate to be presented in national meeting and journal in otolaryngology

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Subjects in this arm will receive pills composed only of Avicel (cellulose filler), starting at 12.5mg nightly, and allowed to increase daily dose by 12.5mg with each subsequent week after enrollment if symptoms not resolved and no adverse effect noted at prior dose, up to maximum dose of 50mg nightly. Treatment duration is 8 weeks
Period: Overall Study
Arm/Group | Amitriptyline | Placebo
Started | 15 | 15
Completed | 10 | 9
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amitriptyline | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 12 | 26
  >=65 years | 1 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (15) | 50 (14) | 48 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 15
  Male | 10 | 5 | 15
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Reflux Symptom Index (RSI) Score [Mean (Standard Deviation); unit: severity on Likert-type scale] | 19 (10) | 24 (10) | 22 (9)

OUTCOME MEASURES:

1. Primary Outcome: Reflux Symptom Index
Description: Reflux symptom index change in score after treatment Range possible: 0 to 45 Higher values indicate worse symptoms / outcomes
Time Frame: 8 weeks
Population: Patients who completed treatment and post-treatment questionnaire
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Amitriptyline | Placebo
Number analyzed (Participants) | 9 | 9
units on a scale | -2.7 (7.1) | 0.3 (12.0)

2. Secondary Outcome: Voice Handicap Index
Description: Voice handicap index change in score after treatment Possible range: 0 to 40 Higher values indicate worse symptoms / outcomes
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Amitriptyline | Placebo
Number analyzed (Participants) | 9 | 9
units on a scale | 3.7 (6.1) | 0 (4.3)

3. Secondary Outcome: Side Effects
Description: number of patients with side effects, type of side effects
Time Frame: 8 weeks
Measure: Number; unit: participants
Groups:
- Amitriptyline: Subjects in this arm will receive pills composed of amitryptline and Avicel (cellulose filler)
  Amitriptyline
- Placebo: Subjects in this arm will receive pills composed only of Avicel (cellulose filler)
  Placebo: Placebo pill
Arm/Group | Amitriptyline | Placebo
Number analyzed (Participants) | 9 | 9
participants
  Dizziness | 4 | 2
  Fatigue | 3 | 1
  Dry mouth | 1 | 2

4. Secondary Outcome: Lost to Follow up
Time Frame: 8 weeks
Population: number of subjects in each arm who were lost to follow up
Measure: Number; unit: participants
Arm/Group | Amitriptyline | Placebo
Number analyzed (Participants) | 15 | 15
participants | 5 | 6

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse event definitions used from http://www.fda.gov/downloads/Drugs/Guidances/ucm073122.pdf, Sections 1.2, 1.50, 1.60; http://www.fda.gov/downloads/Drugs/.../Guidances/UCM227351.pdf
  Full definitions not listed due to character limit of 500
Arm/Group | Amitriptyline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 6/15 | 2/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amitriptyline (N=15) | Placebo (N=15)
Adverse Effect (Nervous system disorders) | 6 (15) | 2 (15) — Not an adverse event. Non-serious adverse effects include dizziness, fatigue, and dry mouth.

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No